CLINICAL TRIAL: NCT03279770
Title: Circulating Non-coding RNAs and Cardiovascular Outcomes in Patients With Dyslipidemia and Atherosclerosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201505165RINC
Record Dates: First submitted 2017-05-11; First posted 2017-09-12 (Actual); Last update posted 2017-09-15 (Actual); Status verified 2017-09

CONDITIONS: Cardiovascular Diseases
Keywords: lnRNA; CV disease
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Plasma and serum Non-coding RNAs
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Cardiovascular diseases and stroke are the major causes of morbidity and death in Taiwan. There is a clear need to identify novel mediators of atherosclerosis in dyslipidemic patients to provide insights into the pathogenesis, to tailor clinical care based on cardiovascular risks, and to develop new therapeutic strategies.

While the roles of lncRNAs in human diseases including cancer and neurodegenerative disorders are beginning to emerge, it remains unclear how lncRNA regulation contributes to atherosclerotic vascular diseases in patients with dyslipidemia. In this proposal, we seek to apply next-generation sequencing technology to investigate circulating (plasma and peripheral blood mononuclear cells [PBMC]) lncRNA expression in control subjects and in dyslipidemic patients with and without atherosclerotic vascular diseases (CAD, ischemic stroke and PAOD). The results from these experiments will lead to better understanding of how circulating lncRNAs contribute to atherosclerotic cardiovascular complications.

DETAILED DESCRIPTION:
Cardiovascular diseases and stroke are the major causes of morbidity and death in Taiwan. Patients with dyslipidemia are prone to atherosclerosis, which predispose to various cardiovascular pathology including coronary artery disease (CAD), ischemic stroke and peripheral artery occlusive disease (PAOD). There are, however, no reliable biomarkers to detect atherosclerotic vascular diseases among dyslipidemic patients or to predict the risks of cardiovascular morbidities and mortality among patients with atherosclerosis. There is a clear need to identify novel mediators of atherosclerosis in dyslipidemic patients to provide insights into the pathogenesis, to tailor clinical care based on cardiovascular risks, and to develop new therapeutic strategies.

It has become increasingly clear that the transcription of the eukaryotic genome is far more pervasive and complex than previously appreciated. While the expression of messenger RNAs (mRNAs) and microRNAs (miRNAs) account for only ~1% of all transcribed species, up to 90% of the mammalian genome is transcribed as long non-coding RNAs (lncRNAs), a heterogeneous group of non-coding transcripts longer than 200 nucleotides. LncRNAs have been shown to be functional and involved in specific physiological and pathological processes through epigenetic, transcriptional and post-transcriptional mechanisms. While the roles of lncRNAs in human diseases including cancer and neurodegenerative disorders are beginning to emerge, it remains unclear how lncRNA regulation contributes to atherosclerotic vascular diseases in patients with dyslipidemia.

In this proposal, we seek to apply next-generation sequencing technology to investigate circulating (plasma and peripheral blood mononuclear cells [PBMC]) lncRNA expression in control subjects and in dyslipidemic patients with and without atherosclerotic vascular diseases (CAD, ischemic stroke and PAOD). We will test the hypothesis that circulating lncRNA expression signature can reflect the atherosclerotic disease states in patients with dyslipidemia. A gene co-expression network analysis will be conducted to identify lncRNAs that are functionally involved in the pathogenesis of atherosclerosis. With the experimental results from an initial dyslipidemic cohort, we will establish an atherosclerosis scoring model on the basis of circulating lncRNA expression signature to facilitate the detection of atherosclerotic vascular diseases in patients with dyslipidemia. The accuracy, sensitivity and specificity of the lncRNA-based atherosclerosis scoring system will then be tested in an independent, large validation cohort. Next, we propose to test the hypothesis that circulating lncRNAs can be novel prognostic biomarkers to predict atherosclerosis progression and cardiovascular outcomes in dyslipidemic patients. The results from these experiments will lead to better understanding of how circulating lncRNAs contribute to atherosclerotic cardiovascular complications. These studies will also establish a set of novel, lncRNA-based diagnostic and prognostic biomarker in dyslipidemic patients to improve clinical preventive and therapeutic care. In addition, the findings from these studies will help to develop novel therapeutic strategies to treat or prevent atherosclerotic vascular diseases in patients with dyslipidemia.

ELIGIBILITY:
Inclusion Criteria:

1. Dyslipidemia: Total cholesterol (TC) >200 mg/dL; LDL-C > 130 mg/dL ; TG > 200 mg/dL; male HDL-C < 40 mg/dL, female HDL-C < 50 mg/dL, or under lipid lowering therapy
2. Atherosclerotic vascular disease:

   1. Coronary atherosclerosis as evidenced by cardiac catheterization examination, having history of myocardial infarction as evidenced by ECG or hospitalization, angina patient showing ischemic ECG changes or positive response to stress test;
   2. Cerebral vascular disease, cerebral infarction, intracerebral hemorrhage (excluding intracerebral hemorrhage associated with other diseases); transient ischemic attack (TIA) with carotid artery ultrasound confirming atheromatous change with more than 70% blockage;
   3. Peripheral atherosclerosis with symptoms of ischemia and confirmed by Doppler ultrasound or angiography in history.
3. Control subjects: Age, gender-matched healthy adults without dyslipidemia and atherosclerotic diseases will be recruited as control subjects.

Exclusion Criteria The main exclusion criteria will be hemodynamically significant valvular or congenital heart disease, life-threatening malignancy, treatment with immunosuppressive agents, or any condition or situation which, in the opinion of the investigator, might be not suitable for this registration.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with dyslipidemia, atherosclerotic vascular diseases, or at least one CV risk factors
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2015-06 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Composite cardiovascular outcome | up to 5 years
  The composite cardiovascular (CV) outcome will be any CV events (coronary, cerebral, or peripheral vascular diseases)

CONTACTS AND LOCATIONS:
Overall Officials: Chau-Chung Wu, M.D., Ph. D., Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes